CLINICAL TRIAL: NCT06563050
Title: Comparison Between Nebulized Lidocaine, Lidocaine Spray, or Their Combination for Topical Anesthesia During Diagnostic Flexible Bronchoscopy: a Randomized Trial
Brief Title: Comparison Between Different Ways for Using Lidocaine During FB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bassem Gadallah Gad-Elkariem Kalam, Resident doctor at Chest Diseases Department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Lidocaine use during FB
Record Dates: First submitted 2024-08-05; First posted 2024-08-20 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Lidocaine Spray; Nebulized Lidocaine; Lung Diseases; Lung Cancer
Keywords: flexible bronchoscopy
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects in group A underwent nebulization with 5 mL of 2% lidocaine for 15 minutes by using a jet nebulizer.
  In group B will underwent 10% lidocaine spray solution will be sprayed 10 times at the oropharynx at 5 s interval.
  Group C: both nebulization and spray will be performed in the same manner except the number of spray will be 2 instead 10.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study subjects will not be blinded; the bronchoscopist and the assessor of outcomes will be blinded to the group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nebulized lidocaine (Experimental): Subjects in group A underwent nebulization with 5 mL of 2% lidocaine for 15 minutes by using a jet nebulizer.
  Interventions: Procedure: Nebulized lidocaine
- Lidocaine spray (Experimental): In group B will underwent 10% lidocaine spray solution will be sprayed 10 times at the oropharynx at 5 s interval.
  Interventions: Procedure: Lidocaine spray
- Combination( Nebulized lidocaine and lidocaine spray) (Experimental): Group C: both nebulization and spray will be performed in the same manner except the number of spray will be 2 instead 10.
  Interventions: Procedure: Combination of nebulized lidocaine and lidocaine spray

INTERVENTIONS:
Procedure: Nebulized lidocaine — Subjects in group A underwent nebulization with 5 mL of 2% lidocaine for 15 minutes by using a jet nebulizer.
  Arms: Nebulized lidocaine
Procedure: Lidocaine spray — Subjects in group B will underwent 10% lidocaine spray solution will be sprayed 10 times at the oropharynx at 5 s interval.
  Arms: Lidocaine spray
Procedure: Combination of nebulized lidocaine and lidocaine spray — Group C: both nebulization and spray will be performed in the same manner except the number of spray will be 2 instead 10.
  Arms: Combination( Nebulized lidocaine and lidocaine spray)

SUMMARY:
compare the efficacy and safety of nebulized lidocaine, oropharyngeal lidocaine spray, or their combination for better outcome of topical anesthesia in subjects undergoing diagnostic FB; severity of cough , pain during procedure , cumulative dose of anesthesia needed and its adverse reaction , overall satisfaction .

DETAILED DESCRIPTION:
Flexible bronchoscopy (FB) is a commonly performed procedure in the diagnosis and treatment of several respiratory disease. Although FB is generally a short procedure, it is uncomfortable for the patient. At least the use of topical anesthesia during FB is essential, especially when performed without sedation. Effective topical anesthesia blunts airway reflexes such as gag, cough, and laryngospasm.

The reduction in cough not only improves patient comfort but also makes the procedure easier for the operator.

Among agents used for topical anesthesia, lidocaine is the most widely used drug because of its safety and favorable pharmacokinetic profile.

Lidocaine is available in various formulations (gel or solution) and can be delivered to the respiratory passages by using different modes (spray, nebulization, transtracheal injection, bronchoscope instillation, and others).

In this study, will compare the efficacy and safety of nebulized lidocaine, oropharyngeal lidocaine spray, or their combination for topical anesthesia in subjects undergoing diagnostic FB, for better outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old will undergo FB are included in this study.

Exclusion Criteria:

* known hypersensitivity to lidocaine.
* Pregnancy.
* hemodynamic instability.
* failure to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The severity of cough using cough severity index | During and within 3 hours after procedure
  Assess the severity of cough during and within 4 hours after the procedure as (0 : absent cough is better ) , ( 5 : disturbing cough is the worst )
pain during the procedure rated by the subjects on the Faces Pain Rating Scale. | During and within 3 hours after procedure
  As (0 : no pain , the best) , ( 10 : worst pain )
time taken to cross the vocal cords. | at the beginning of the procedure(time zero) till seconds after crossing the vocal cords
  the median time in seconds will be calculated during the procedure from the introduction the tip of bronchoscope from the nostril to second at which the tip of bronchoscopy cross the the vocal cords.
changes in heart rate | During and within 3 hours after procedure
  changes in the heart rate from the baseline before procedure
Changes in oxygen saturation | During and within 3 hours after procedure
  changes in the oxygen saturation from the baseline before procedure

SECONDARY OUTCOMES:
cumulative dose of lidocaine administered during the procedure. | During the procedure
  Less cumulative dose of lidocaine needed during the procedure is better
adverse reactions to lidocaine | During and within 3 hours after procedure
  assess for any adverse effects related to lidocaine use especially arrhythmia or other adverse effects as convulsions, involuntary movements, bronchospasm, and anaphylaxis.
overall satisfaction with the procedure using likert scale . | During and within 3 hours after procedure
  As (1 : strongly disagree , is the worst) and (5 : strongly agree , is better)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mostafa Abdelhadi, Study Director — Professor of Chest Diseases and Tuberculosis; Montaser Gamal Ahmed, Study Director — lecturer of Chest Diseases and Tuberculosis; Nermeen Mohammed Abuelkassem, Study Director — lecturer of Chest Diseases and Tuberculosis

IPD SHARING:
Plan to Share IPD: Yes